CLINICAL TRIAL: NCT02857491
Title: Comparison of Intravitreal Injection of Ranibizumab Versus Sham Injection Before Vitrectomy in Patients With Proliferative Diabetic Retinopathy: a Single-center, Prospective Double-blinded Randomized Controlled Trial
Brief Title: Intravitreal Injection of Ranibizumab Versus Sham Before Vitrectomy in Patients With Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, Director of Fundus Disease Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014MEKY034
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid; Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ranibizumab (Experimental): Intravitreal Injection of 0.5 mg ranibizumabone week before vitrectomy.
  Interventions: Drug: ranibizumab; Procedure: pars plana vitrectomy
- control (Sham Comparator): Sham intravitreal injection one week before vitrectomy.
  Interventions: Drug: sham; Procedure: pars plana vitrectomy

INTERVENTIONS:
Drug: ranibizumab — intravitreal injection of 0.5 mg ranibizumab before vitrectomy
  Other Names: Lucentis
  Arms: ranibizumab
Drug: sham — sham intravitreal injection before vitrectomy
  Other Names: control
  Arms: control
Procedure: pars plana vitrectomy — surgical procedure to remove the intravitreal hemorrhage and fibrosis membrane, and re-attach the retina, and perform endo laser photocoagulation on retina.
  Other Names: vitrectomy

SUMMARY:
Certain percent of the eyes with proliferative diabetic retinopathymay require pars plana vitrectomy (PPV) due to vitreous haemorrhage, proliferative membrane, and tractional retinal detachment. This study will compare intravitreal injection of anti-vascular endothelial growth factor (ranibizumab) versus sham injection before vitrectomy for PDR. The main focus is to see if pre-operative injection of ranibizuman can reduce peri-operative hemorrahge related complications.

DETAILED DESCRIPTION:
Eyes responding to panretinal photocoagulation can remain stable for decades, but incomplete responses and relapses can occur in a certain percent of diabetic patients showing as proliferative diabetic retinopathy. At present vitrectomy is the main intervention for those eyes with vitreous hemorrhage, proliferative membrane, and tractional retinal detachment. And the surgical procedure might be complicated because of intraoperative bleeding. And post-operative complications might be also involved. Perioperative use of intraocular anti-VEGF might be associated with less hemorrhage related complications and better visula acuity. This study will compare intravitreal injection of anti-vascular endothelial growth factor (ranibizumab) versus sham injection one week before surgery. The investigators tried to make sure whether pre-operative injection of ranibizuman can reduce reduce intra-operative bleeding, reduce the frequency of using endodiathermy, decrease surgical time, improve microcurculation of retina, and elevte best-corrected visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* type I or type II diabetes
* there is clear indications for vitrectomy due to proliferative membrane in the vitreoretinal interface, mild hemorrhage, or tractional retinal detachment
* retinal large vessels could be detected within one PD away from the edge of optic disc by OCT
* microcurculation could be detected by FFA in at least one quadrant
* the patient could tolerant FFA examination

Exclusion Criteria:

* a history of vitrectomy or scleral bucke in the included eye
* retinal laser photocoagulation treatment within 90 days in the included eye
* anti-VEGF treatment with 90 days in either eye
* there is cocurrent neovascular glaucoma in the included eye
* any reason that might hinde the procedure of vitrectomy, FFA OCT or the observation of ocular fudus
* a history of cere-brovascular accident or heart stroke
* renal failure
* could not attend follow up regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
perioperative hemorrhage of the surgical eye | 3 month

SECONDARY OUTCOMES:
size of retinal non-perfusion area assessed by fluorescene angiography | 3 month
macular retinal thickness assessed with optical coherance tomography | 3 month
retinal vessel oxygen saturation measured with a retinal oximeter | 3 months
best-corrected visual acuity | 3 months

OTHER OUTCOMES:
complications | 3 months
  other perioperative complications
surgical time | 1 day
grade of surgical difficulty | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No